CLINICAL TRIAL: NCT00772356
Title: A Monocenter, Open-Label Glucose Clamp Study Examining the Metabolic Effect of Insulin Infusion Intervals for Basal Insulin Infusion in Patients With Type I Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000559; 05/0377-Basal
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- A (Experimental)
  Interventions: Device: Accu-Chek Spirit Insulin Pump
- B (Active Comparator)
  Interventions: Device: Comparator insulin pump

INTERVENTIONS:
Device: Accu-Chek Spirit Insulin Pump
  Arms: A
Device: Comparator insulin pump
  Arms: B

SUMMARY:
This crossover, glucose-clamp study will investigate the impact of different basal insulin infusion rates on glucose control employing insulin pumps with different insulin delivery regimen. Patients will be randomized in one of 2 groups, to receive on the first study day insulin via pumps with pulsatile or quasi-continuous delivery modes. On the second study day they will be switched to treatment with the alternative delivery regimen. The anticipated duration of the trial is 2 study days and the target sample size is 14 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18-65 years of age
* Type I diabetes mellitus
* Currently on continuous subcutaneous insulin infusion therapy

Exclusion Criteria:

* Proliferative retinopathy or maculopathy requiring actue treatment within last 6 months
* Use of systemic corticoids in last 3 months
* Treatment with medication known to interfere with glucose metabolism

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Comparison of glucose infusion rate necessary to keep blood glucose constant | Throughout study

SECONDARY OUTCOMES:
Serum insulin and free fatty acid levels | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Dr. Petersen, Study Director — Roche Diagnostics GmbH
Locations (1):
- Neuss, Germany